CLINICAL TRIAL: NCT04519970
Title: (COMEBACK): Biktarvy in PLWH But Not Retained in Care Coupled With a Strengths-based Case Management Approach to Assess Virologic Suppression Rates and Retention in Care, Along With Patient Reported Outcomes (PROS).
Brief Title: Clinical Opportunities and Management to Exploit Biktarvy as Asynchronous Connection Key (COMEBACK)
Acronym: COMEBACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gregory Huhn (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Gregory Huhn, MD, MPHTM Attending Physician, Ruth M. Rothstein CORE Center
Organization: Ruth M. Rothstein CORE Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IN-US-380-5725
Record Dates: First submitted 2020-08-10; First posted 2020-08-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-08

CONDITIONS: Hiv
Keywords: Adherence; Case Management; Biktarvy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Highest Tier of Case Management (Piggyback) and Biktarvy (Active Comparator): The most intensive tier of case management. Includes three appointment reminders; check ins twice per week; travel compensation; housing support; food insecurity support; follow ups for missed appointments and off pill counts; connections with substance use programs; meetings with the benefits department for health insurance needs; childcare support to make appointments; mental healthcare referrals; open pool appointments as back-up options in case of rescheduling needs; late doctor's appointments and prescription pick up for those working during the day; meetings with the health educators to discuss HIV and ART; and re-motivation of HIV treatment every 3 months.
  Interventions: Behavioral: Case Management
- Middle Tier of Case Management (Got Your Back) and Biktarvy (Active Comparator): The middle tier (Got Your Back) will work closely with the CORE case managers to augment their work in housing support, transportation assistance, mental healthcare referrals, childcare assistance, substance use program referrals, food insecurity support and health insurance needs. The retention specialist will additionally provide this middle tier 2 reminders for appointments; check ins once per week; follow ups for missed appointments or off pill counts; support with scheduling appointments for limited availability; meetings with the health educators for information on HIV or ART; and re-motivation for treatment at the 6 and 9 month marks of participation.
  Interventions: Behavioral: Case Management
- Lowest Tier of Case Management (Backbone) and Biktarvy (Active Comparator): The top tier (Backbone) will need the least amount of support and also have a CORE Center case manager for a majority of the support in housing, food, insurance, transportation, childcare, substance use, and mental healthcare. The retention specialist will still provide an appointment reminder; check ins every other week; text checkups after missed appointments or off pill counts; support with scheduling for appointments or prescription pick up for limited availability; and re-motivation of treatment for HIV at the 9 month mark of study participation.
  Interventions: Behavioral: Case Management

INTERVENTIONS:
Behavioral: Case Management — Each tier will have a different level of case management and support, all with the goal of increasing adherence to Biktarvy for HIV management.

SUMMARY:
COMEBACK is an investigator-initiated, 48-week study. The study will be conducted in 100 persons living with HIV (PLWH) who have been off ART for two or more weeks. All enrolled participants will be prescribed Biktarvy, if determined appropriate upon review of past historical resistance tests, for use throughout the study period. Participants will also complete a series of Patient Reported Outcomes (PROs) at screening and be assigned one of three tiers of case management intervention (Piggyback, Got Your Back, Backbone), with each tier increasing in intensity regarding intervention techniques and options provided. Participants will be assessed for virologic suppression, retention in care, and PROS throughout study follow up and at study end.

DETAILED DESCRIPTION:
In most settings in the US when patients out of care and off of ART reengage with clinical providers routine labs are collected, including CMP, CD4, VL, and HIV resistance testing when indicated, healthcare benefits are reassessed, and the most recent ART regimen is restarted if the patient agrees to treatment. There may be characteristics of these regimens that may present barriers to sufficient adherence, or perform suboptimally in patients with certain immunologic and/or viral factors, which may impact virologic suppression, including multiple pills, drug-drug interactions, variable tolerability, low CD4, high VL, or low thresholds for resistance. Biktarvy is a Single Tablet Regimen (STR) with high potency and good tolerability that can be safely used in multiple patient groups, with features, including activity in patients with a history of multi-class resistance, that may facilitate immediate ART reinitiation among a broad population of patients reengaging in care in order to promote rapid virologic suppression. Addressing this important patient population with poor retention with support mechanisms to reengage in care and reinitiate effective ART immediately may improve retention in care and accelerate virologic suppression as likewise derived in immediate ART models in treatment-naïve patients, and represent a touchstone to drive sustainability in preventing new HIV transmissions in a high burden area to meet the goals of reducing HIV as a public health threat over the next 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected
2. Not on ART for >2 weeks
3. History of estimated eGFR > 30 ml3/min
4. Baseline labs (CBC, CMP, CD4+, HIV-1 RNA) and resistance genotype test collected <2 weeks or on day of Biktarvy ART reinitiation
5. 18 years or older

Exclusion Criteria:

1. No history of primary integrase inhibitor mutations, >3 TAMs, K70E, Q151M, T69 insertion, or K65R + M184V/I on prior resistance testing
2. Drug-drug interactions with Biktarvy
3. Pregnancy
4. Unable or unwilling to provide consent for study participation
5. Any condition that, in the opinion of the Investigator of Record (IoR), would make participation in the study unsafe, complicate interpretation of outcome data, or otherwise interfere with achieving the study objective.
6. Current participation in another ART adherence study
7. Allergy to bictegravir, emtricitabine or tenofovir alafenamide
8. Signs or symptoms of opportunistic infection with cryptococcal meningitis, tuberculosis or other infection that requires delay of reinitiation of antiretroviral therapy
9. Concomitant use of medications that are contraindicated with bictegravir, emtricitabine and tenofovir alafenamide including adefovir, carbamazepine, cladribine, dofetilide, fosphenytoin-phenytoin, oxcarbazepine, phenobarbital, primidone, rifampin, rifabutin, rifapentine, St. John's Wort, tipranavir

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2024-04-06 (Actual)

PRIMARY OUTCOMES:
Virologic Suppression Rates | 1 year
  Number of patients with virologic suppression, defined as HIV RNA <200 copies/ml at week 48 RNA.
Retention in Care | 1 year
  Number of patients retained in study, defined as at least 2 visits or 2 HIV-1 RNA viral load reports occurring at least 3 months apart within the 12-month study time period

SECONDARY OUTCOMES:
Patient Reported Outcomes concerning social and health related barriers | 1 year
  Favorable outcomes concerning health and and social related determinants as assessed by responses to a series of Patient Reported Outcomes at 6 and 12 months. See full list in attached documents.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Huhn, MD, MPHTM, Principal Investigator — Ruth M. Rothstein CORE Center
Locations (1):
- Ruth M. Rothstein CORE Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No